CLINICAL TRIAL: NCT06796452
Title: Effect of First and Second Rib Mobilization on Pain, Range of Motion, Muscle Endurance and Disability in Patients With Non-Specific Neck Pain
Brief Title: Effect of First and Second Rib Mobilization in Patients With Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0156
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain; Mobilization
Keywords: Cervical ribs; Endurance
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ribs Mobilization (Experimental): will receive Maitland first and second Rib Mobilization with three sets of 6-8 repetitions in each session and conventional(Baseline) Physical therapy Treatment.
  Interventions: Other: Ribs Mobilization
- Conventional Treatment (Active Comparator): will only receive Baseline Physical therapy treatment
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Ribs Mobilization — Three sets of 6-8 repetitions in each session and conventional(Baseline) Physical therapy Treatment.
  Arms: Ribs Mobilization
Other: Conventional treatment — * Hot pack for 8 min
  * Maitland Generalized Cervical Mobilizations (6-8 REPS,3 sets)
  * Isometric Strengthening Exercise
  Arms: Conventional Treatment

SUMMARY:
This study will be a randomized controlled trial.Non-probability convenient sampling will be used to collect the data. Sample size of 44 subjects with age group between 20-45 years will be taken. Data will be collected from the patients having present complaint of nonspecific Neck pain. Outcome measures will be taken using Numeric pain rating scale (NPRS) for pain, Neck Disability Index (NDI), Muscle endurance by Muscle endurance test using stopwatch and Universal Goniometer (GU) for Range of motion. An informed consent will be taken. Subjects will be selected on the basis of inclusion and exclusion criteria and will be equally divided into two groups by random computer generated numbers method. Group A will receive first and second rib mobilization, and Group B will receive conventional treatment. Outcome measures will be measured prior and after 4 weeks. Data will be analyzed by SPSS version 25.

DETAILED DESCRIPTION:
the effect of First Rib Mobilization in Mechanical Neck Pain with Radiculopathy for Pain Relief in which fifty patients with age between 21- 60 years, who fulfilled the study sample selection criteria were registered in the study. After sample selection of 50 subjects (by scientific calculator) by using convenient sampling technique, a written consent was signed from each participant before any assessment and management. All subjects were treated by applying Maitland grade I, II first rib mobilization for a session comprising on 20 minutes. The subjects were treated thrice in a week for next 2 weeks. The participants were assessed before and after treatment. Numeric Pain Rating Scale (NPRS) was used to record pain severity level. A self-structured validated questionnaire was used to collect the demographics. Pain was assessed before and after first rib mobilization by using paired sample t-test was done to see the changes in the mean pain score. The study concluded that First Rib Mobilization was an effective treatment for subjects with mechanical neck ache and radicular symptoms.

Despite the extensive research on non-specific neck pain (NSNP) and various therapeutic interventions, there is a notable gap in the literature regarding the specific effects of first and second rib mobilization on pain, range of motion, muscle endurance, and disability in patients with NSNP. While studies have explored manual therapies, proprioceptive exercises, and virtual reality as complementary interventions, the direct impact of rib mobilization, especially involving both the first and second ribs, remains under-investigated. Additionally, most existing studies focus on short-term outcomes, and there is limited evidence on the long-term effects of rib mobilization techniques.

ELIGIBILITY:
Inclusion Criteria:

* Neurological tests will be negative
* Both genders having age between 20 to 45 years
* Participants should have primary complaint of neck pain
* Neck Disability Index (NDI) score of 20% or greater (i.e. 10 points or greater on a 0 to 50 scale)
* a pain intensity of ≥4 on the 10-point Numerical Pain Rating Scale (NPRS)

Exclusion Criteria:

* First and second rib fracture and dislocation
* Past surgical history of cervical and thoracic region
* Thoracic Outlet syndrome and Cervical radiculopathy
* Congenital anomalies of spine and ribs

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-13 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | 4 weeks
  Patient level of pain will be assessed using this scale by interview method. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain".
Universal Goniometer | 4 weeks
  The range of motion will be measured using universal goniometer

SECONDARY OUTCOMES:
Muscle Endurance Test using Stopwatch | 4 weeks
  Muscle endurance of neck extensors and flexors will be measured by using stopwatch for readings
Neck Disability Index | 4 weeks
  Neck disability will be assessed using this scale. The Neck Disability Index (NDI) scores disability on a scale of 0 to 50, with 0 representing no disability and 50 representing complete disability. A score can also be converted to a percentage by doubling it. Here's a breakdown of the scoring and interpretation:
  0-4 points (0-8%): No disability. 5-14 points (10-28%): Mild disability. 15-24 points (30-48%): Moderate disability. 25-34 points (50-64%): Severe disability. 35-50 points (70-100%): Complete disability. The NDI consists of 10 questions, each scored from 0 to 5, with higher numbers indicating a higher self-reported disability. The total score is the sum of the scores from each question

CONTACTS AND LOCATIONS:
Overall Officials: Syed Sramad Hussain Bukhari, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Murtaza Rehabilitation center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No